CLINICAL TRIAL: NCT04871854
Title: Comparative Study Evaluating Clinical Outcomes for Patients Treated With Tocilizumab for Sever COVID-19 Infection in Breast Cancer Patients Versus Non Cancer Patients
Brief Title: Evaluating Tocilizumab for Sever COVID-19 Infection in Breast Cancer vs. Non Cancer Pateints
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, ALshaimaa Ibrahim Rabie, Assistant lecturer , pharm D, October 6 University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-H-PHBSU-21010
Record Dates: First submitted 2021-04-25; First posted 2021-05-04 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — tocilizumab; Absorptiometry, Photon

STUDY DESIGN:
Intervention Model Description: comparative study two Covid-19 infected groups selected according to preexisting sever Covid -19 patients receiving Tocilizumab versus traditional thherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Svere infected Covid-19 control (Experimental): Arm one confirmed sever COVID 19 infection admitted to ICU including with or without breast cancer patients comorbidity receive traditional therapy
  Interventions: Drug: traditional Covid -19 therapy
- sever infected Covid -19 pateints study (Active Comparator): Arm two patients with confirmed sever COVID 19 infection admitted to ICU with or without breast cancer patients comorbidity tocilizumab
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — patients treated with Tocilizumab for Covid-19 infection
  Other Names: Actemra
  Arms: sever infected Covid -19 pateints study
Drug: traditional Covid -19 therapy — patients treated with traditional therapy for Covid-19 infection
  Other Names: DExa /Corticosteriods
  Arms: Svere infected Covid-19 control

SUMMARY:
To compare evaluating Clinical outcomes for patients treated with with or without breast cancer patients comorbidity for sever COVID-19 infection in breast cancer patients versus non cancer patients and evaluating Tocilizumab efficacy versus traditional therapy

DETAILED DESCRIPTION:
Cancer patients considered to be one of the least population that can be considered lucky during COVID 19 pandemic attributed that to long term treatment with chemotherapy, immunosuppression and multi comorbidities . Women with breast cancer are more likely to get covid-19 infection rather than other type cancers . the co-existing of two diseases breast cancer and Covid19 are very challengeable due to confusion and similarities found in clinical biomarkers to evaluate both diseases as ferritin, D dimers and C-reactive protein and all other immune response and cytokine storm syndrome especially including interleukin-6 (IL-6) . using chemotherapy or any other cytotoxic drugs may exacerbate the severity of COVID -19 infection as well as poor clinical outcomes and even death are expected . The anti-human IL-6R monoclonal antibody (Tocilizumab) was used first in China in patients with severe COVID-19 and patients improved in different clinical outcome . In cancer patients particularly the issue is debatable about the benefits of receiving Tocilizumab.

Clinical studies are going on such medication role in treatment of patients with severe covid 19 infection however, studies have not clearly addressed the role of Tocilizumab breast cancer patient compared to non-cancer patients. This study aims to measure different clinical outcomes after using Tocilizumab in sever covid 19 infection in breast cancer patients vs. non cancer patients

ELIGIBILITY:
Inclusion Criteria:

1. patients admitted to ICU with or without breast cancer (non-metastatic) comorbidity
2. age 18-85 years' old
3. moderate to sever confirmed COVID 19 infection through PCR and CT
4. male or female
5. confirmed Covid-19 by PCR
6. Requiring ICU admission
7. WITH evidence of severe COVID-19 (at least 2 of the following):

   1. Fever > 38C within 72 hours
   2. Pulmonary infiltrate on chest X ray /ground glass opacity
   3. Need for supplemental O2 to maintain saturation > 92%
8. AND at least 1 of the following:

   1. Ferritin > 500 ng/ml
   2. CRP > 50 mg/L
   3. LDH >250 U/L
   4. D-dimer > 1000 ng/mL
9. all patient assigned informed consent

Exclusion Criteria:

1. above 85 years' old
2. metatastic breast cancer
3. autoimmune disease patients
4. Unable to provide verbal informed consent
5. preganncy
6. Subjects between the ages of 70 and 75 will be excluded if they have NYHA Class III/IV heart failure
7. Active TB
8. Receipt of IV tocilizumab for the treatment of a non-COVID condition within 3 weeks of the first COVID symptom
9. History of hypersensitivity to tocilizumab 7. ANC <500, Platelets <50,000* 8. AST/ALT > 5X ULN

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) after treatment of Tocilizumab | 28 days time fram
  measure mortality rate
progression free survival (PFS) | 3 months
  measure time from recovery until reinfection with Covid-19 after treatment of Tocilizumab
time of improvement or worsening at least one point change in ordinal scale | 28 days
  Time to improvement will be assessed by changes on the clinical improvement or worsening as it measures illness severity over time ,by using Ordinal Scale for Clinical Improvement which score zero indicate no clinical or evidence virologic infection and high score 8 indicate death

SECONDARY OUTCOMES:
measure percentage of patients need Mechanical Ventilation Required (Including CPAP) during Follow up period, Supplemental Oxygen required | 28 days time fram
  complications
Duration of mechanical ventilation | 28 days
  Duration of mechanical ventilation from the start to end
adverse effect | 28 days
  any side effects or serious adverse effect
length of stay in Intensive care unit | 28 days
  admission date and discharge date documented and LOS calculated from the day of admission to day of discharge, and based on the number of nights spent in hospital. Patients admitted and discharged on the same day have a length of stay of less than one day. dividing the sum of inpatient days by the number of patients admissions.

CONTACTS AND LOCATIONS:
Overall Officials: Raghda Hussein, PHD, Study Director — Beni suef university fculty of pharmacy; Ahmed Hassan shaaban, MD, Study Director — clinical oncology faculty of medicine Beni suef university; Doaa Mahmoud, MD, Principal Investigator — Beni-Suef University
Locations (1):
- ALsafwa specialized hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No